CLINICAL TRIAL: NCT05431023
Title: Efficacy of Lactoferrin as Adjunct Therapy for Pneumonia in Children and Adolescents
Brief Title: Effect of Lactoferrin in Pneumonia Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Omima mahran hussein, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pneumonia
Record Dates: First submitted 2022-03-12; First posted 2022-06-24 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia | interventions — Lactoferrin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with pneumonia who receive only treatment for pneumonia (Experimental): They receive only treatment for pneumonia
  Interventions: Drug: Pneumonia treatment
- pneumonia patients receive treatment for pneumonia and lactoferrin (Experimental): They receive treatment for pneumonia and lactoferrin
  Interventions: Drug: Lactoferrin; Drug: Pneumonia treatment

INTERVENTIONS:
Drug: Lactoferrin — Lactoferrin binds to and blocks glycosaminoglycan viral receptors, especially heparan sulfate (HS). The binding of LF and HS prevents the first contact between virus and host cell and therefore prevents the infection
  Arms: pneumonia patients receive treatment for pneumonia and lactoferrin
Drug: Pneumonia treatment — Antibiotics for pneumonia

SUMMARY:
Pneumonia is defind as the inflammation of lung tissue caused by an infectious agent that results in acute respiratory signs and symptoms. Community acquired pneumonia (CAP) is a major cause of morbidity and increased health care costs. In developing nations, pneumonia remains a significant cause of mortality in children.

Pneumonia occurs in 30 to 45 of every 1,000 children under 5 years of age; it is less common in 5- to 9-year olds (16 to 22/1,000) and in older children (7 to 16/1,000).

Streptococcus pneumoniae is the primary bacterial cause of pneumonia in infants and children. Viral etiologies become less prevalent and mycoplasmal and chlamydial infections become more prevalent with increasing age

DETAILED DESCRIPTION:
Lactoferrin (LF) is iron-binding glycoprotein of the transferrin family that is expressed and secreted by glandular cells and is found in most body fluids . It appears at especially high concentrations in mammalian milk and was first identified in bovine milk , and was subsequently isolated from human milk.

LFs bacteriostatic function is due to its ability to take up the Fe3+ ion, limiting use of this nutrient by bacteria at the infection site and inhibiting the growth of these microorganisms as well as the expression of their virulence factors .

ELIGIBILITY:
Inclusion Criteria:

* Pneumonia patients
* from the age of one month to the age of 18 years .

Exclusion Criteria:

Neonates and any children with :

* immune deficiency
* congenital heart disease
* neuromascular disorder
* genetic syndromes

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Survival rate. | Up to 8 weeks
  Comparing the influence of the intervention on the Survival rate.

SECONDARY OUTCOMES:
Mean change in the disease severity (clinical assessment) | Up to 4 weeks
  Recording the changes from severe to moderate or mild and the time taken